CLINICAL TRIAL: NCT03093402
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Multicenter Study to Evaluate Efficacy, Safety, and Tolerability of JBT-101 in Systemic Lupus Erythematosus
Brief Title: JBT-101 in Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Corbus Pharmaceuticals Inc. (Industry); Autoimmunity Centers of Excellence (Other); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT ALE09; NIAID CRMS ID#: 30147 (Other: DAIT NIAID); UM1AI110494 (NIH)
Record Dates: First submitted 2017-02-21; First posted 2017-03-28 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Systemic Lupus Erythematosus; SLE; Lupus
Keywords: JBT-101 (also known as lenabasum); efficacy; musculoskeletal disease; randomized trial
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Musculoskeletal Diseases | interventions — lenabasum; anabasum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JBT-101: 5 mg Twice Daily (Experimental): Eligible subjects will receive assigned study treatment of JBT-101 5 mg administered twice daily.
  Interventions: Drug: JBT-101
- JBT-101: 20 mg & Placebo (Experimental): Eligible subjects will receive assigned study treatment of JBT-101 20 mg (A.M. Study Product) and 20 mg Placebo (P.M. Study Product).
  Interventions: Drug: JBT-101; Drug: Placebo
- JBT-101: 20 mg Twice Daily (Experimental): Eligible subjects will receive assigned study treatment of JBT-101 20 mg (A.M. Study Product) and JBT-101 20 mg (P.M. Study Product).
  Interventions: Drug: JBT-101
- Placebo + Placebo (Placebo Comparator): Eligible subjects will receive assigned study treatment of Placebo (A.M.) and Placebo (P.M.) for (JBT-101).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JBT-101 — Participants will self-administer JBT-101 by mouth (orally), at prescribed dose and frequency per protocol, Days 1-84. Administration of dose(s) should be at least 8 hours apart.
  Other Names: lenabasum; anabasum; resunab; ajulemic acid; CT-3; IP751; CPL7075
  Arms: JBT-101: 20 mg & Placebo; JBT-101: 20 mg Twice Daily; JBT-101: 5 mg Twice Daily
Drug: Placebo — Participants will self-administer JBT-101 placebo by mouth (orally), at prescribed dose and frequency per protocol, Days 1-84. Administration of dose(s) should be at least 8 hours apart.
  Other Names: JBT-101 placebo; lenabasum placebo
  Arms: JBT-101: 20 mg & Placebo; Placebo + Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety, and tolerability of JBT-101 (also known as lenabasum) in systemic lupus erythematosus (SLE).

* One hundred adults with active joint disease and at least moderate pain will be enrolled in this study to evaluate treatment of their systemic lupus erythematosus (SLE) with JBT-101. JBT-101 is a synthetic endocannabinoid receptor type 2 (CB2) agonist and an activator of the body's normal processes, to resolve innate immune responses without immunosuppression.
* Participants will receive 2 doses of JBT-101 by mouth (three groups of varying doses) or, placebo, for 84 days and will continue to be followed for an additional 28 days. Participant visits to assess endpoints occur on Day 1, then every 2 weeks twice, then every 4 weeks three times, for a total of six visits.
* The change in maximum daily pain Numerical Rating Scale (NRS) score from Baseline (Visit 1) will be assessed at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills the updated American College of Rheumatology (ACR) 1982 Revised Criteria for the Classification of Systemic Lupus Erythematosus;
* At least 3 months of treatment with an anti-malarial drug such as hydroxychloroquine or a history of intolerance, contraindication, or unwillingness to take an anti-malarial drug;
* Meets the Safety of Estrogen in Lupus: National Assessment (SELENA) Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) definition of arthritis (Petri et al., 1999) or mild/moderate arthritis or tendonitis scored as a BILAG B on the updated BILAG 2004;
* Seven-day average of maximum of daily pain Numerical Rating Scale (NRS) scores ≥ 4 out of 10;
* Overlap with polymyositis, systemic sclerosis, Sjögren's syndrome, or rheumatoid arthritis is allowed, if, in the site investigator's judgment, the predominant clinical features are those of Systemic Lupus Erythematosus (SLE);
* Not expected by the site investigator to require a change in potential disease- modifying treatments for SLE from Screening through Visit 6 (Day 112);
* Willing to not start nor stop any Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) or potential disease-modifying medications or supplements for SLE from Screening through Visit 6 (Day 112), unless a change is recommended by the site investigator or other treating physicians;
* Willing not to use any legal or illegal cannabinoids, including Food and Drug Administration (FDA)-approved cannabinoids or cannabinoid-mimic drugs, or any illegal substance of abuse from Screening through Visit 6 (Day 112);
* If a woman of child-bearing potential, willing to use one of the highly effective (failure rate < 1% per year) birth control method from Screening through Visit 6 (Day 112) or for 28 ± 3 days after the last dose of study product; and
* Willing to follow instructions, complete study procedures and attend study visits as required by this protocol.

Exclusion Criteria:

* Severe or unstable Systemic lupus erythematosus (SLE), such as any one of the following:

  * A British Isles Lupus Activity Group (BILAG) A score in one or more BILAG domains at Screening;
  * Treatment with any intraarticular, intravenous, or intramuscular systemic corticosteroids within 14 days of Screening;
  * Treatment with oral prednisone > 10 mg per day or > 20 mg every other day (or equivalent dose of another corticosteroid) within 14 days of Screening;
  * Increased dose of systemic corticosteroids in the 14 days prior to Screening;
  * Treatment with cyclophosphamide or anti-TNFalpha biologic agents within 3 months before Visit 1 (Day 1);
  * Treatment with B cell-depleting monoclonal antibodies (rituximab, Ocrelizumab, anti-CD22) within 6 months before Visit 1 (Day 1);
  * Treatment with methotrexate, mycophenolate, azathioprine, leflunomide, cyclosporine, belimumab, tacrolimus, or any other immunosuppressive agent not included in 2b.-d. above, when the dose of that immunosuppressive agent has increased within 3 months before Visit 1. Concurrent treatment with any of these medications is allowed as long as the doses have been stable for at least 3 months before Visit 1 (Day 1); or
  * Actively listed on an organ transplantation list or have received an organ transplant other than a corneal transplant.
* Significant diseases or conditions other than SLE that may influence response to the study product or safety, such as:

  * Active bacterial or viral infection requiring systemic antibiotic or anti-viral treatment within 14 days before Visit 1 (Day 1);
  * Acute or chronic hepatitis B or C infection;
  * Human immunodeficiency infection (HIV);
  * History of active tuberculosis or positive tuberculosis skin or blood test without: 1) completing a course of appropriate treatment; or ) having received at least one month of appropriate treatment prior to Visit 1 (Day 1) and continuing to receive appropriate treatment during the study;
  * No elective surgery should be planned from Visit 1 (Day 1) through Visit 6 (Day 112); or
  * A history of cancer except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy greater than one year before Visit 1 (Day 1).
  * Significant heart disease as defined by:

    * Uncontrollable congestive heart failure, unstable angina, unstable atherosclerotic cardiovascular disease, significant arrhythmia requiring chronic therapy, pulmonary arterial hypertension with dyspnea, disability rated as New York heart Association Grade III or higher, severe systemic hypertension or severe peripheral vascular disease;
    * Marked baseline prolongation of QT/QTc interval (i.e. repeated demonstration of a QTc interval ≥ 450 msec for males and ≥470 msec for females);
    * History of risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT/QTc syndrome); or
    * Clinically significant confirmed abnormality, as determined by the site investigator or qualified designee, on 12-lead Electrocardiogram (ECG) at Screening or Visit 1 (Day 1) before dosing.
* History of chronic pain requiring treatment with narcotic analgesia for more than 14 days total within 6 months of baseline. This does not include self-limited pain associated with identifiable events such as surgery;
* Current evidence of alcohol abuse (defined as 4 or more drinks per day on at least 4 days of the week) or history of abuse of illegal and/or legally prescribed drugs such as barbiturates, benzodiazepines, amphetamines, cocaine, or opioids during the 1 year prior to Screening;
* Currently pregnant, breast-feeding, or lactating;
* Any investigational agent within 30 days or five therapeutic half-lives of that agent whichever is longer, before Visit 1 (Day 1);
* Any of the following values for laboratory tests at Screening:

  * A positive pregnancy test (also at Visit 1);
  * A newly positive QuantiFERON(R) blood test for tuberculosis, without: 1) completing a course of appropriate treatment; or ) having received at least one month of appropriate treatment prior to Visit 1 and continuing to receive appropriate treatment during the study. If the subject has a previous documented positive tuberculosis skin, then this testing does not need to be repeated. If the subject has a documented negative test result within the last year, testing does not need to be repeated, at the discretion of the site investigator.
  * Hemoglobin < 8 g/dL;
  * Neutrophils < 1.0 x 10^9/L;
  * Platelets < 75 x 10^9/L;
  * Estimated Glomerular Filtration Rate (eGFR) < 50 ml/min according to Cockcroft-Gault equation;
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase > 2.0 x upper limit of normal; or
  * Total bilirubin ≥ 1.5 x upper limit of normal.
* Any other conditions that, in the opinion of the site investigator, are clinically significant and may put the subject at greater safety risk, influence response to study product, or interfere with study assessments. When in doubt, the site investigator or qualified designee should discuss the situation with the Protocol Chairs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meggan Mackay, M.D., M.S., Study Chair — Northwell Health; Robert B. Zurier, M.D., Study Chair — Northwell Health
Locations (16):
- United States (16):
  - University of California San Diego School of Medicine: Division of Rheumatology, Allergy and Immunology, La Jolla, California
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - University of California San Francisco School of Medicine: Lupus Clinic and Rheumatology Clinical Research Center, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Emory University: Division of Rheumatology, Atlanta, Georgia
  - Feinstein Institute for Medical Research: Center for Autoimmune and Musculoskeletal Diseases, Manhasset, New York
  - New York University Langone Medical Center: Department of Medicine, Division of Rheumatology, New York, New York
  - Columbia University Medical Center: Department of Medicine, Division of Rheumatology, New York, New York
  - Bronx-Lebanon Hospital Center: Division of Rheumatology, The Bronx, New York
  - Duke University, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Penn State MS Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center: Division of Rheumatology and Clinical Immunology, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data in ImmPort [https://immport.niaid.nih.gov/ ], a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts, upon completion of the study.
Time Frame: After completion of the study.
Access Criteria: Data is available to the public once Individual Participant-Level data is posted to ImmPort.
URL: http://www.immport.org/

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Autoimmunity Centers of Excellence (ACE) website — http://www.autoimmunitycenters.org/
- See also: Corbus Pharmaceuticals and Clinical Programs in Systemic Lupus Erythematosus — https://www.corbuspharma.com/our-pipeline/endocannabinoid-system

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 study sites were activated in the United States, beginning in December 2017. A total of 148 participants were screened from January 2018 to March 2021 at all 16 sites. 109 participants were randomized.
Groups:
- High: JBT-101 20mg/20mg: Participants self-administered 20 mg of JBT-101 by mouth (orally), twice a day, on Days 1-84.
- Medium: JBT-101 20mg/Placebo: Participants self-administered 20 mg of JBT-101 by mouth (orally), in the morning and Placebo in the evening, on Days 1-84.
- Low: JBT-101 5mg/5mg: Participants self-administered 5 mg of JBT-101 by mouth (orally), twice a day, on Days 1-84.
- Placebo: Participants self-administered Placebo by mouth (orally), twice a day, on Days 1-84.
Period: Overall Study
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Started | 27 | 28 | 26 | 28
Completed | 20 | 23 | 24 | 24
Not Completed | 7 | 5 | 2 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 0 | 1
Not completed — Withdrew prior to dosing | 2 | 1 | 2 | 3
Not completed — Ineligible for study | 1 | 0 | 0 | 0
Not completed — Prescribed a prohibited concomitant medication | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The modified-intent-to-treat population includes all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 24 | 25 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 27 | 23 | 25 | 98
  >=65 years | 2 | 0 | 1 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (12.5) | 40.3 (8.6) | 43.4 (12.6) | 44.6 (9.5) | 44.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 23 | 23 | 95
  Male | 0 | 3 | 1 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 6 | 6 | 25
  Not Hispanic or Latino | 18 | 20 | 18 | 19 | 75
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 9 | 8 | 32
  White | 14 | 15 | 8 | 14 | 51
  More than one race | 1 | 2 | 2 | 1 | 6
  Unknown or Not Reported | 2 | 3 | 3 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 25 | 27 | 24 | 25 | 101
Duration of Systemic Lupus Erythematosus [Mean (Standard Deviation); unit: years] — Duration of Systemic Lupus Erythematosus (SLE) is the number of years at the screening visit since the onset of SLE.
  years | 11.6 (8.3) | 13.1 (10.1) | 10.7 (7.4) | 11.9 (10.9) | 11.9 (9.2)
Screening Fibromyalgia Symptom Scale Score [Mean (Standard Deviation); unit: Scores on a Scale] — The possible score range is from 0 to 31 , with a higher score corresponding to a greater level of symptom severity.
  Scores on a Scale | 16.8 (6.1) | 15.2 (6.2) | 14.2 (6.0) | 16.6 (6.3) | 15.7 (6.2)
Screening Fibromyalgia Symptom Scale Score, Categorical [Count of Participants; unit: Participants]
  <13 | 7 | 8 | 7 | 7 | 29
  >=13 | 18 | 19 | 17 | 18 | 72
Screening 7-day Average Pain NRS [Mean (Standard Deviation); unit: Score] — The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
  Score | 6.6 (1.4) | 6.7 (1.7) | 6.6 (1.4) | 6.5 (1.5) | 6.6 (1.5)
Screening 7-day Average Pain NRS, Categorical [Count of Participants; unit: Participants] — The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
  Participants
    <=6 | 12 | 14 | 12 | 12 | 50
    >6 | 13 | 13 | 12 | 13 | 51
Baseline 7-Day Average Pain NRS [Mean (Standard Deviation); unit: Score] — The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
  Score | 6.6 (1.4) | 6.7 (1.7) | 6.6 (1.6) | 6.6 (1.6) | 6.6 (1.6)
Baseline 7-Day Average Maximum Daily Pain NRS, Categorical [Count of Participants; unit: Participants] — The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
  Participants
    <4 | 0 | 0 | 1 | 0 | 1
    >=4 | 25 | 27 | 23 | 25 | 100
SELENA-SLEDAI Score [Mean (Standard Deviation); unit: Scores on a Scale] — The Safety of Estrogen in Lupus National Assessment (SELENA) Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a validated tool for assessing SLE disease activity. The SLEDAI is a one page assessment that contains 24 items scored as present or absent. Each item is assigned a weighted score which is summed to calculate the overall SLEDAI score. SLEDAI score ranges from 0-105 points. Higher scores represent more disease activity with a score of 6 being considered clinically important and may impact the decision to treat.
  Scores on a Scale | 6.9 (2.7) | 7.0 (2.7) | 7.5 (2.0) | 8.2 (2.3) | 7.4 (2.5)
Arthritis Present on SLEDAI [Count of Participants; unit: Participants] — On the SLEDAI assessment arthritis is defined as > 2 joints with pain and signs of inflammation (i.e., tenderness, swelling, or effusion).
  Participants
    Present | 23 | 24 | 23 | 25 | 95
    Not Present | 2 | 3 | 1 | 0 | 6
Number of Swollen Joints [Mean (Standard Deviation); unit: units on a scale] — Swollen Joint Count (SJC) is calculated based on swelling response of 66joints examined. SJC possible values range from 0 to 66. A lower SJC indicates less joint swelling.
  units on a scale | 5.4 (5.2) | 7.6 (8.7) | 6.8 (6.6) | 9.0 (8.4) | 7.2 (7.4)
Number of Tender Joints [Mean (Standard Deviation); unit: units on a scale] — Tender Joint Count (TJC) is calculated based on tenderness response of 68 joints examined. TJC possible values range from 0 to 68. A lower TJC indicates less joint tenderness.
  units on a scale | 14.1 (11.8) | 15.0 (16.1) | 13.1 (9.6) | 18.4 (10.0) | 15.2 (12.3)
Number of Tender and Swollen Joints [Mean (Standard Deviation); unit: units on a scale] — Tender and Swollen Joint Count is calculated based on both tenderness and swelling response of 66 joints examined. The possible values range from 0 to 66. A lower count indicates less joint tenderness and swelling.
  units on a scale | 4.1 (4.1) | 6.3 (7.8) | 6.5 (6.7) | 8.3 (8.5) | 6.3 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the Maximum Daily NRS-Pain Score at Day 84
Description: The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
  Participants will be asked to report their maximum daily pain using the NRS-Pain. Participants will call into an interactive voice response e diary system (IVRS) and record the number that best reflects their maximum amount of pain experienced in the last 24 hours. Participants will be asked to call at the same time each day, preferably before bedtime.
  Longitudinal trends over the course of the treatment period will be modeled and used to estimate difference between means at baseline and Day 84 for each treatment group.
Time Frame: Day 1 through Day 84
Population: The modified intent-to-treat population includes all randomized participants who received at least one dose of study drug. One participant, in the Medium: JBT-101 20mg/Placebo treatment, took one dose of drug in clinic and subsequently decided to discontinue treatment and terminate the study. This participant did not report a pain NRS score on Day 1 and is therefore not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: NRS Pain Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 26 | 24 | 25
NRS Pain Score
  Day 1 | 6.3 [5.9 to 6.7] | 6.4 [6.0 to 6.8] | 6.0 [5.6 to 6.4] | 6.2 [5.7 to 6.7]
  Day 84 | 5.1 [4.1 to 6.1] | 4.9 [4.0 to 5.8] | 5.1 [4.1 to 6.0] | 5.9 [4.8 to 7.0]
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The null hypothesis is that linear trends from Day 1 to Day 84 are equivalent for each active JBT-101 cohort and placebo. The overall test is a 3 degree of freedom F test that simultaneously compares the estimated mean change from Day 1 to Day 84 for each of the 3 active JBT-101 cohorts versus placebo; Test type: Superiority — The fixed effects included treatment, time, time² , time- and time² by treatment interactions. The Screening FSS score and the Screening 7-day average maximum daily pain NRS were included as covariates. Within-subject random effects for intercept and slopes for time and time² were fit using an unstructured covariance matrix, assuming a different structure for placebo and pooled active treatment groups; p = 0.4190, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the estimated mean change from Day 1 to Day 84 for each of the 3 active treatment arms versus placebo; Median Difference (Final Values) = -0.9, 95% CI 2-sided [-2.5 to 0.6] — Mean difference in the change from Day 1 to Day 84 for High JBT-101 - Placebo. The estimated mean change (95% confidence interval) from Day 1 to Day 84 for Placebo was -0.3 (-1.5, 0.9)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4190, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Median Difference (Final Values) = -1.2, 95% CI 2-sided [-2.7 to 0.3] — Mean difference in the change from Day 1 to Day 84 for Medium JBT-101 - Placebo. The estimated mean change (95% confidence interval) from Day 1 to Day 84 for Placebo was -0.3 (-1.5, 0.9)
Statistical Analysis 3: Comparison: Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.4190, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-2.2 to 0.8] — Mean difference in the change from Day 1 to Day 84 for Low JBT-101 - Placebo. The estimated mean change (95% confidence interval) from Day 1 to Day 84 for Placebo was -0.3 (-1.5, 0.9)

2. Secondary Outcome: Number of Participants With No Pain, Mild Pain, Moderate Pain or Severe Pain in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
Time Frame: Visit 1 (Baseline)
Population: The modified intent-to-treat population includes all randomized participants who received at least one dose of study drug and had data at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Participants
  No Pain | 0 | 0 | 0 | 0
  Mild Pain | 0 | 0 | 0 | 0
  Moderate Pain | 14 | 18 | 14 | 16
  Severe Pain | 11 | 9 | 10 | 9

3. Secondary Outcome: Number of Participants With No Pain, Mild Pain, Moderate Pain or Severe Pain in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: as for outcome 2
Time Frame: Visit 3 (Day 29)
Population: The modified intent-to-treat population includes all randomized participants who received at least one dose of study drug and had data at Visit 3 (Day 29).
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 21 | 24 | 23 | 25
Participants
  No Pain | 0 | 0 | 0 | 1
  Mild Pain | 3 | 3 | 5 | 0
  Moderate Pain | 14 | 16 | 12 | 17
  Severe Pain | 4 | 5 | 6 | 7

4. Secondary Outcome: Number of Participants With No Pain, Mild Pain, Moderate Pain or Severe Pain in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: as for outcome 2
Time Frame: Visit 4 (Day 57)
Population: The modified intent-to-treat population includes all randomized participants who received at least one dose of study drug and had data at Visit 4 (Day 57).
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 18 | 23 | 22 | 23
Participants
  No Pain | 2 | 2 | 0 | 0
  Mild Pain | 2 | 1 | 4 | 3
  Moderate Pain | 11 | 16 | 13 | 14
  Severe Pain | 3 | 4 | 5 | 6

5. Secondary Outcome: Number of Participants With No Pain, Mild Pain, Moderate Pain or Severe Pain in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: as for outcome 2
Time Frame: Visit 5 (Day 85)
Population: The modified intent-to-treat population includes all randomized participants who received at least one dose of study drug and had data at Visit 5 (Day 85).
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 19 | 21 | 22 | 22
Participants
  No Pain | 0 | 1 | 1 | 0
  Mild Pain | 5 | 4 | 4 | 1
  Moderate Pain | 12 | 12 | 13 | 15
  Severe Pain | 2 | 4 | 4 | 6

6. Secondary Outcome: Number of Participants With No Pain, Mild Pain, Moderate Pain or Severe Pain in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: as for outcome 2
Time Frame: Visit 6 (Day 113)
Population: The modified intent-to-treat population includes all randomized participants who received at least one dose of study drug and had data at Visit 6 (Day 113).
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 11 | 16 | 15 | 11
Participants
  No Pain | 0 | 1 | 0 | 0
  Mild Pain | 1 | 2 | 5 | 0
  Moderate Pain | 8 | 10 | 9 | 9
  Severe Pain | 2 | 3 | 1 | 2

7. Secondary Outcome: Change From Baseline in the Improvement Pain Category Prior to Study Visits
Description: The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain. The Improvement Pain Category is the change in the pain category from baseline to the post-baseline visit. An improvement of at least 2 pain categories from baseline is considered major pain improvement; improvement of 1 pain category, improvement; no change in pain category, no change; worsening of at least 1 pain category, worsening.
Time Frame: Visit 3 (Day 29)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 21 | 24 | 23 | 25
Participants
  Major Improvement | 1 | 1 | 1 | 1
  Improvement | 7 | 5 | 7 | 3
  No Change | 13 | 18 | 14 | 20
  Worsening | 0 | 0 | 1 | 1

8. Secondary Outcome: Change From Baseline in the Improvement Pain Category Prior to Study Visits
Description: as for outcome 7
Time Frame: Visit 4 (Day 57)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 18 | 23 | 22 | 23
Participants
  Major Improvement | 2 | 2 | 0 | 0
  Improvement | 5 | 5 | 9 | 6
  No Change | 10 | 16 | 12 | 17
  Worsening | 1 | 0 | 1 | 0

9. Secondary Outcome: Change From Baseline in the Improvement Pain Category Prior to Study Visits
Description: as for outcome 7
Time Frame: Visit 5 (Day 85)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 19 | 21 | 22 | 22
Participants
  Major Improvement | 2 | 1 | 2 | 1
  Improvement | 7 | 7 | 8 | 2
  No Change | 10 | 13 | 11 | 19
  Worsening | 0 | 0 | 1 | 0

10. Secondary Outcome: Change From Baseline in the Improvement Pain Category Prior to Study Visits
Description: as for outcome 7
Time Frame: Visit 6 (Day 113)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 11 | 16 | 15 | 11
Participants
  Major Improvement | 0 | 1 | 1 | 0
  Improvement | 4 | 5 | 7 | 4
  No Change | 6 | 9 | 7 | 7
  Worsening | 1 | 1 | 0 | 0

11. Secondary Outcome: Percentage of Participants Who Had at Least 30% Improvement From Baseline in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: The numeric rating scale for pain (NRS-Pain) consists of an 11-point NRS ranging from 0 (no pain) to 10 (pain as bad as you can imagine). A rating of 1-3 is considered mild pain; 4-6, moderate pain; and 7-10, severe pain.
  The percent change from baseline in the 7-day average of the maximum NRS-Pain scores prior to study Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85 - Last Day of Treatment) and Visit 6 (Day 113)
Population: mITT: The number analyzed is mITT with available data at each visit. Due to dropout or missing scores, not everyone in mITT has data to contribute at each visit
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Participants
  Day 29: number analyzed (Participants) | 21 | 24 | 23 | 25
  Day 29 | 19.0 | 33.3 | 30.4 | 20.0
  Day 57: number analyzed (Participants) | 18 | 23 | 22 | 23
  Day 57 | 38.9 | 47.8 | 40.9 | 26.1
  Day 85: number analyzed (Participants) | 19 | 21 | 22 | 22
  Day 85 | 42.1 | 42.9 | 40.9 | 27.3
  Day 113: number analyzed (Participants) | 11 | 16 | 15 | 11
  Day 113 | 36.4 | 31.3 | 46.7 | 27.3
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each active treatment vs. placebo at Day 29; Test type: Superiority; p = 0.594, Mixed Models Analysis
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each active treatment vs. placebo at Day 57; Test type: Superiority; p = 0.487, Mixed Models Analysis
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each active treatment vs. placebo at Day 85; Test type: Superiority; p = 0.760, Mixed Models Analysis
Statistical Analysis 4: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each active treatment vs. placebo at Day 113; Test type: Superiority; p = 0.676, Mixed Models Analysis

12. Secondary Outcome: Percentage of Participants Who Had at Least 50% Improvement From Baseline in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: as for outcome 11
Time Frame: as for outcome 11
Population: mITT - The number analyzed is mITT with available data at each visit. Due to dropout or missing scores, not everyone in mITT has data to contribute at each visit
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Participants
  Day 29: number analyzed (Participants) | 21 | 24 | 23 | 25
  Day 29 | 14.3 | 16.7 | 17.4 | 8.0
  Day 57: number analyzed (Participants) | 18 | 23 | 22 | 23
  Day 57 | 16.7 | 13.0 | 18.2 | 13.0
  Day 85: number analyzed (Participants) | 19 | 21 | 22 | 22
  Day 85 | 26.3 | 23.8 | 22.7 | 4.5
  Day 113: number analyzed (Participants) | 11 | 16 | 15 | 11
  Day 113 | 9.1 | 12.5 | 20.0 | 0
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.796, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 29 testing that the proportion of subjects with >= 50% improvement is equal among the 4 treatment groups
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.955, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 57 testing that the proportion of subjects with >= 50% improvement is equal among the 4 treatment groups
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.211, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 85 testing that the proportion of subjects with >= 50% improvement is equal among the 4 treatment groups
Statistical Analysis 4: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.481, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 113 testing that the proportion of subjects with >= 50% improvement is equal among the 4 treatment groups

13. Secondary Outcome: Percentage of Participants Who Had at Least 75% Improvement From Baseline in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits Score
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Participants
  Day 29: number analyzed (Participants) | 21 | 24 | 23 | 25
  Day 29 | 0 | 4.2 | 8.7 | 4.0
  Day 57: number analyzed (Participants) | 18 | 23 | 22 | 23
  Day 57 | 11.1 | 8.7 | 4.5 | 4.3
  Day 85: number analyzed (Participants) | 19 | 21 | 22 | 22
  Day 85 | 5.3 | 4.8 | 9.1 | 0
  Day 113: number analyzed (Participants) | 11 | 16 | 15 | 11
  Day 113 | 0 | 12.5 | 0 | 0
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.790, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 29 testing that the proportion of subjects with >= 75% improvement is equal among the 4 treatment groups
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.843, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 57 testing that the proportion of subjects with >= 75% improvement is equal among the 4 treatment groups
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.637, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 85 testing that the proportion of subjects with >= 75% improvement is equal among the 4 treatment groups
Statistical Analysis 4: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.243, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 113 testing that the proportion of subjects with >= 75% improvement is equal among the 4 treatment groups

14. Secondary Outcome: Percentage of Participants Who Had 100% Improvement From Baseline in the 7-day Average of the Maximum NRS-Pain Score Prior to Study Visits
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Participants
  Day 29: number analyzed (Participants) | 21 | 24 | 23 | 25
  Day 29 | 0 | 0 | 0 | 0
  Day 57: number analyzed (Participants) | 18 | 23 | 22 | 23
  Day 57 | 0 | 4.3 | 0 | 0
  Day 85: number analyzed (Participants) | 19 | 21 | 22 | 22
  Day 85 | 0 | 4.8 | 4.5 | 0
  Day 113: number analyzed (Participants) | 11 | 16 | 15 | 11
  Day 113 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; JBT-101 High, JBT-101 Medium, JBT-101 Low, Placebo; Test type: Superiority; p > 0.999, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 57 testing that the proportion of subjects with >=100% improvement is equal among the 4 treatment groups
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; JBT-101 High, JBT-101 Medium, JBT-101 Low, Placebo; Test type: Superiority; p = 0.861, Exact Likelihood Ratio Test — This p-value is from an exact likelihood ratio test at Day 85 testing that the proportion of subjects with >= 100% improvement is equal among the 4 treatment groups

15. Secondary Outcome: Change From Baseline in Physician Assessed Tender Joint Count
Description: The change from baseline in the number of tender joints identified by the physician in the Physician Joint Exam at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed. The number of tender joints can range from 0 to 68 joints.
Time Frame: Baseline, (Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Number of Tender Joints
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Number of Tender Joints
  Baseline/ Day 1 | 14.1 (11.8) | 15.0 (16.1) | 13.1 (9.6) | 18.4 (10.0)
  Day 29: number analyzed (Participants) | 20 | 24 | 24 | 24
  Day 29 | 12.1 (13.3) | 12.3 (18.5) | 8.8 (9.3) | 10.0 (9.0)
  Day 57: number analyzed (Participants) | 19 | 22 | 24 | 23
  Day 57 | 9.5 (10.5) | 12.3 (20.2) | 5.0 (6.9) | 10.7 (12.1)
  Day 85: number analyzed (Participants) | 19 | 22 | 23 | 22
  Day 85 | 10.3 (13.8) | 11.9 (20.2) | 4.7 (6.0) | 11.3 (11.8)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.390, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline tender joint count at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-4.8 to 8.7] — Mean difference in the change from baseline tender joint count for High JBT-101 - Placebo. The estimated tender joint count mean change from baseline (95% confidence interval) for Placebo was -6.3 (-12.0, -0.7)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.390, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]; Mean Difference (Final Values) = 1.7, 95% CI 2-sided [-4.9 to 8.2] — Mean difference in the change from baseline tender joint count for Medium JBT-101 - Placebo. The estimated tender joint count mean change from baseline (95% confidence interval) for Placebo was -6.3 (-12.0, -0.7)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.390, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]; Median Difference (Final Values) = -2.0, 95% CI 2-sided [-8.6 to 4.6] — Mean difference in the change from baseline tender joint count for Low JBT-101 - Placebo. The estimated tender joint count mean change from baseline (95% confidence interval) for Placebo was -6.3 (-12.0, -0.7)

16. Secondary Outcome: Change From Baseline in Physician Assessed Swollen Joint Count
Description: The change from baseline in the number of swollen joints identified by the physician in the Physician Joint Exam at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed. The number of swollen joints can range from 0 to 66 joints.
Time Frame: Baseline, (Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Number of Swollen Joints
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Number of Swollen Joints
  Baseline/ Day 1 | 5.4 (5.2) | 7.6 (8.7) | 6.8 (6.6) | 9.0 (8.4)
  Day 29: number analyzed (Participants) | 20 | 24 | 24 | 24
  Day 29 | 5.6 (8.5) | 4.0 (5.0) | 4.5 (7.2) | 5.3 (7.0)
  Day 57: number analyzed (Participants) | 19 | 22 | 24 | 23
  Day 57 | 3.4 (5.1) | 3.0 (4.7) | 2.3 (2.8) | 5.1 (5.7)
  Day 85: number analyzed (Participants) | 19 | 22 | 23 | 22
  Day 85 | 3.3 (5.7) | 3.1 (5.7) | 2.1 (3.0) | 4.0 (4.1)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.556, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline swollen joint count at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Median Difference (Final Values) = 0.7, 95% CI 2-sided [-1.6 to 3.0] — Mean difference in the change from baseline swollen joint count for High JBT-101 - Placebo. The estimated swollen joint count mean change from baseline (95% confidence interval) for Placebo was -4.0 (-5.7, -2.4)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.556, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline swollen joint count at Day 85 for each JBT-101 cohort versus placebo; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.5 to 2.0] — Mean difference in the change from baseline swollen joint count for Medium JBT-101 - Placebo. The estimated swollen joint count mean change from baseline (95% confidence interval) for Placebo was -4.0 (-5.7, -2.4)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.556, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-3.1 to 1.4] — [estimate comment as in outcome 16, analysis 1]

17. Secondary Outcome: Percentage of Participants With Presence of Arthritis in SELENA-SLEDAI
Description: The Safety of Estrogen in Lupus National Assessment (SELENA) Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a validated tool for assessing SLE disease activity.
  The percentage of participants with arthritis indicated as Present on the SELENA SLEDAI at Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed. [A single question on the SELENA SLEDAI with a response of Present or Absent was assessed.]
Time Frame: as for outcome 11
Population: mITT - The number analyzed is mITT with available data at each visit. Due to dropout or missing scores, not everyone in mITT has data to contribute at each visit."
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Participants
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 14.3 | 28.0 | 20.8 | 16.0
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 30.0 | 39.1 | 45.8 | 25.0
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 45.0 | 39.1 | 47.8 | 33.3
  Day 113: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 113 | 15.0 | 39.1 | 34.8 | 25.0
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 29; Test type: Superiority; p = 0.669, Mixed Models Analysis
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 57; Test type: Superiority; p = 0.432, Mixed Models Analysis
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 85; Test type: Superiority; p = 0.780, Mixed Models Analysis
Statistical Analysis 4: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 113; Test type: Superiority; p = 0.285, Mixed Models Analysis

18. Secondary Outcome: Percentage of Participants With Improvement From Baseline in Arthritis in BILAG-2004
Description: The BILAG-2004* is a validated index for assessing SLE disease activity. The BILAG-2004 includes 97 clinical and laboratory items to evaluate SLE disease activity in 9 organ systems. The severity of arthritis at baseline will be determine by the highest arthritis severity level where arthritis is indicated as improving, same, new or worse* BILAG-2004: British Isles Lupus Assessment Group 2004. The percentage of participants who met the criteria for improvement of arthritis in the BILAG-2004 Musculoskeletal assessments (using the mild, moderate and severe arthritis questions on the assessment) at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Number; unit: Percentage of Subjects
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 23 | 24
Percentage of Subjects | 50.0 | 56.5 | 78.2 | 58.3

19. Secondary Outcome: Percentage of Participants as Responders Using the SLE Responder Index (SRI)
Description: The SRI is a validated SLE disease activity instrument used to detect clinically meaningful improvement of disease in SLE clinical trials. The SRI is a composite instrument comprised of the SELENA-SLE Disease Activity Index [SELENA-SLEDAI], Physician Global Assessment (PGA) and British Isles Lupus Assessment Group (BILAG) 2004. A responder is defined as having at least a 4 point reduction in the SELENA-SLEDAI score, no new BILAG A or no more than 1 new BILAG B domain score, and no increase in the PGA of 0.3 points or more. The percentage of participants who met the criteria for a responder in the SRI at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Number; unit: Percentage of Subjects
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Subjects
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 19.0 | 28.0 | 25.0 | 20.0
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 40.0 | 34.8 | 41.7 | 33.3
  Day 85: number analyzed (Participants) | 20 | 23 | 22 | 23
  Day 85 | 50.0 | 39.1 | 54.5 | 39.1
  Day 113: number analyzed (Participants) | 19 | 23 | 21 | 24
  Day 113 | 21.1 | 34.8 | 33.3 | 29.2
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; JBT-101 High, JBT-101 Medium, JBT-101 Low, Placebo; Test type: Superiority — The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 29; p = 0.872, Mixed Models Analysis
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; JBT-101 High, JBT-101 Medium, JBT-101 Low, Placebo; Test type: Superiority — The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 57; p = 0.895, Mixed Models Analysis
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; JBT-101 High, JBT-101 Medium, JBT-101 Low, Placebo; Test type: Superiority — The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 85; p = 0.669, Mixed Models Analysis
Statistical Analysis 4: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; JBT-101 High, JBT-101 Medium, JBT-101 Low, Placebo; Test type: Superiority — The dichotomous outcome is modeled using the generalized estimating equations approach under the binomial distribution with a logit link. The model includes fixed effects for visit, treatment and visit*treatment interaction with an unstructured within-subject correlation structure across visits. The overall test p-value is a 3 degree-of-freedom test comparing each of the 3 active treatments vs. placebo at Day 113; p = 0.668, Mixed Models Analysis

20. Secondary Outcome: Change From Baseline in Lupus Disease Activity - SELENA-SLEDAI Score
Description: The change from baseline in the SELENA-SLEDAI score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
  The Safety of Estrogen in Lupus National Assessment (SELENA) Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a validated tool for assessing SLE disease activity. The SLEDAI is a one page assessment that contains 24 items scored as present or absent. Each item is assigned a weighted score which is summed to calculate the overall SLEDAI score. SLEDAI score ranges from 0-105 points. Higher scores represent more disease activity, with a score of 6 being considered clinically important and may impact the decision to treat.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: mITT -The number analyzed is mITT with available data at each visit. Due to dropout or missing scores, not everyone in mITT has data to contribute at each visit
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Scores on a Scale
  Baseline/Day 1 | 6.9 (2.7) | 7.0 (2.7) | 7.5 (2.0) | 8.2 (2.3)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 6.1 (2.2) | 5.5 (3.2) | 6.0 (2.9) | 6.6 (3.2)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 5.4 (3.4) | 4.5 (2.6) | 5.0 (3.2) | 6.1 (3.3)
  Day 85: number analyzed (Participants) | 20 | 23 | 22 | 23
  Day 85 | 4.7 (3.0) | 4.5 (2.4) | 4.5 (3.1) | 5.5 (3.6)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = .820, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline SELENA-SLEDAI Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.3 to 1.5] — Mean difference in the change from baseline SLEDAI score for High JBT-101 - Placebo. The estimated Day 85 SLEDAI mean change from baseline (95% confidence interval) for Placebo was -2.2 (-3.6, -0.8)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = .820, Mixed Models Analysis — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.0 to 1.8] — Mean difference in the change from baseline SLEDAI score for Medium JBT-101 - Placebo. The estimated Day 85 SLEDAI mean change from baseline (95% confidence interval) for Placebo was -2.2 (-3.6, -0.8)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = .820, Mixed Models Analysis — [p-value comment as in outcome 20, analysis 1]; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.6 to 1.1] — Mean difference in the change from baseline SLEDAI score for Low JBT-101 - Placebo. The estimated Day 85 SLEDAI mean change from baseline (95% confidence interval) for Placebo was -2.2 (-3.6, -0.8)

21. Secondary Outcome: Change From Baseline in Lupus Disease Activity - Total BILAG-2004 Score
Description: For each of the nine domains, a numerical score will be assigned based on the BILAG score as follows: A=12, B=8, C=1 and D/E=0. A single numerical BILAG total score will be calculated for each participant visit as the summation of the numerical scores for each of the nine domains. The BILAG total score can range from 0 to 108, with higher scores indicating more disease activity. The change from baseline in the total BILAG-2004 score at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed. The BILAG-2004* is a validated index for assessing SLE disease activity. The BILAG-2004 includes 97 clinical and laboratory items to evaluate SLE disease activity in 9 organ systems.
  * BILAG-2004: British Isles Lupus Assessment Group 2004.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1: number analyzed (Participants) | 24 | 27 | 23 | 24
  Baseline/Day 1 | 12.2 (5.8) | 9.7 (4.8) | 11.5 (3.6) | 13.1 (4.3)
  Day 29: number analyzed (Participants) | 21 | 25 | 23 | 24
  Day 29 | 8.8 (5.9) | 5.8 (4.9) | 6.2 (4.3) | 5.5 (4.3)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 23
  Day 57 | 7.9 (6.4) | 6.5 (5.5) | 5.4 (4.8) | 8.1 (5.6)
  Day 85: number analyzed (Participants) | 18 | 23 | 21 | 22
  Day 85 | 8.6 (5.6) | 5.1 (5.1) | 4.9 (5.0) | 7.7 (6.2)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = .244, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline BILAG total score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-3.0 to 4.4] — Mean difference in the change from baseline BILAG score for High JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -4.3 (-7.0, -1.5)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = .244, Mixed Models Analysis — [p-value comment as in outcome 21, analysis 1]; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-5.2 to 2.0] — Mean difference in the change from baseline BILAG score for Medium JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -4.3 (-7.0, -1.5)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = .244, Mixed Models Analysis — [p-value comment as in outcome 21, analysis 1]; Median Difference (Final Values) = -2.6, 95% CI 2-sided [-6.2 to 0.9] — Mean difference in the change from baseline BILAG score for Low JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -4.3 (-7.0, -1.5)

22. Secondary Outcome: Change From Baseline in Lupus Disease Activity -Physician's Global Assessment (PGA) Score
Description: The change from baseline in the total PGA score at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed. The PGA utilizes a 0 to 3 visual analogue scale for assessing disease activity in SLE that is anchored by the verbal descriptors as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe. An increase of >=0.3 points is considered worsening of the PGA.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1 | 1.2 (0.6) | 1.2 (0.5) | 1.4 (0.4) | 1.3 (0.5)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 1.2 (0.6) | 0.9 (0.6) | 1.0 (0.6) | 1.1 (0.5)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 1.0 (0.5) | 0.8 (0.5) | 0.9 (0.5) | 1.0 (0.6)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 0.9 (0.5) | 0.8 (0.5) | 0.7 (0.5) | 0.9 (0.6)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.408, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline Physician's Global Assessment (PGA) Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.27 to 0.40] — Mean difference in the change from baseline PGA score for High JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -0.43 (-0.70, -0.15)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.408, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 1]; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.40 to 0.26] — [estimate comment as in outcome 22, analysis 1]
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.408, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.50 to 0.16] — Mean difference in the change from baseline PGA score for Low JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -0.43 (-0.70, -0.15)

23. Secondary Outcome: Change From Baseline in Lupus Disease Activity- Patient Global Assessment Score
Description: The change from baseline in the total Patient Global Assessment score at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed. The total Patient Global Assessment is performed with a visual analogue scale (0 to 100) in which the participant is asked to indicate how active she/he thinks their disease is. The visual analogue scale is anchored by two descriptors: "not active" (score of 0) and "extremely active" (score of 100).
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1: number analyzed (Participants) | 25 | 27 | 24 | 24
  Baseline/Day 1 | 60.2 (22.4) | 67.0 (22.1) | 65.6 (20.5) | 65.5 (15.0)
  Day 29: number analyzed (Participants) | 20 | 23 | 23 | 23
  Day 29 | 48.1 (27.6) | 49.2 (29.1) | 47.5 (31.7) | 54.4 (21.7)
  Day 57: number analyzed (Participants) | 18 | 23 | 24 | 23
  Day 57 | 48.3 (24.0) | 50.5 (29.6) | 50.2 (28.2) | 59.4 (26.0)
  Day 85: number analyzed (Participants) | 19 | 23 | 23 | 21
  Day 85 | 37.0 (24.8) | 48.0 (26.2) | 48.7 (30.0) | 58.7 (22.7)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.070, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline Patient Global Assessment Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -21.48, 95% CI 2-sided [-37.24 to -5.72] — Mean difference in the change from baseline Patient Global Assessment score for High JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -5.27 (-16.11, 5.56)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.070, Mixed Models Analysis — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Final Values) = -10.40, 95% CI 2-sided [-25.33 to 4.54] — [estimate comment as in outcome 23, analysis 1]
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.070, Mixed Models Analysis — [p-value comment as in outcome 23, analysis 1]; Mean Difference (Final Values) = -10.81, 95% CI 2-sided [-25.78 to 4.16] — Mean difference in the change from baseline Patient Global Assessment score for Low JBT-101 - Placebo. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -5.27 (-16.11, 5.56)

24. Secondary Outcome: Change in Baseline in PROMIS-29 Short Form Score - Physical Function T-score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Short Form (Version 2.0) will be used to assess trends over time in this state of health measure. The PROMIS-29 consists of 7 domains related to physical, mental and social health. Raw scores are calculated for each domain and translated into a T-score per the PROMIS-29 scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents better functioning for the Physical Function domain.
  The change from baseline in the PROMIS-29 Physical Function T-score at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85).
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
T-Score
  Baseline/Day 1 | 37.7 (6.4) | 39.2 (8.3) | 39.2 (6.0) | 38.5 (4.4)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 38.5 (7.7) | 39.8 (6.1) | 42.1 (7.8) | 40.5 (8.0)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 39.9 (8.2) | 40.0 (7.7) | 42.2 (7.8) | 40.4 (7.6)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 39.8 (8.7) | 41.1 (7.4) | 41.5 (7.7) | 40.3 (7.0)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.979, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline Physical Function T-score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Median Difference (Final Values) = 0.30, 95% CI 2-sided [-3.38 to 3.99] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 1.8 (-0.8, 4.3)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.979, Mixed Models Analysis — [p-value comment as in outcome 24, analysis 1]; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [-3.13 to 3.93] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 1.8 (-0.8, 4.3)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.979, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Physical Function Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Median Difference (Final Values) = 0.77, 95% CI 2-sided [-2.77 to 4.31] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was 1.8 (-0.8, 4.3)

25. Secondary Outcome: Change in Baseline in PROMIS - Anxiety T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Anxiety T-Score will be used to assess trends over time in this health measure.
  The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents worse symptomology for the Anxiety domain. The change from baseline in PROMIS Anxiety Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
T-Score
  Baseline/Day 1 | 57.0 (8.6) | 52.4 (10.2) | 56.9 (9.8) | 55.1 (11.4)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 54.7 (11.2) | 53.2 (10.3) | 54.1 (7.5) | 51.6 (11.1)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 55.7 (10.0) | 52.6 (11.4) | 56.0 (9.9) | 53.4 (10.8)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 52.9 (10.1) | 50.0 (8.5) | 54.7 (9.2) | 53.5 (10.6)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.788, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Anxiety T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -1.44, 95% CI 2-sided [-6.14 to 3.26] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -1.8 (-4.8, 1.2)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.788, Mixed Models Analysis — [p-value comment as in outcome 25, analysis 1]; Mean Difference (Final Values) = -1.56, 95% CI 2-sided [-6.07 to 2.96] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -1.8 (-4.8, 1.2)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.788, Mixed Models Analysis — [p-value comment as in outcome 25, analysis 1]; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-4.00 to 4.94] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -1.8 (-4.8, 1.2)

26. Secondary Outcome: Change in Baseline in PROMIS - Depression T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Depression T-Score will be used to assess trends over time in this health measure. The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents worse symptomology for the Depression domain. The change from baseline in PROMIS Depression Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1 | 57.7 (10.2) | 49.6 (10.1) | 52.7 (8.8) | 52.1 (10.0)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 53.8 (11.5) | 49.1 (9.6) | 49.8 (7.9) | 52.0 (10.9)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 52.9 (10.6) | 49.7 (10.4) | 51.8 (9.1) | 51.1 (10.9)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 53.0 (10.6) | 50.0 (9.2) | 50.0 (7.9) | 50.6 (10.4)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.766, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Depression T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -1.49, 95% CI 2-sided [-6.14 to 3.16] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -1.7(-4.6, 1.3)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.766, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Final Values) = 0.76, 95% CI 2-sided [-3.60 to 5.11] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -1.7(-4.6, 1.3)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.766, Mixed Models Analysis — [p-value comment as in outcome 26, analysis 1]; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-5.55 to 3.07] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -1.7(-4.6, 1.3)

27. Secondary Outcome: Change in Baseline in PROMIS - Fatigue T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Fatigue T-Score will be used to assess trends over time in this health measure. The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents worse symptomology for the Fatigue domain. The change from baseline in PROMIS Fatigue Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
T-Score
  Baseline/Day 1 | 64.0 (7.1) | 62.4 (11.9) | 63.1 (9.9) | 63.7 (9.7)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 61.8 (9.6) | 59.6 (11.4) | 58.0 (11.4) | 60.1 (13.4)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 61.7 (9.2) | 57.8 (11.3) | 55.8 (10.6) | 59.4 (11.6)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 59.7 (11.0) | 56.7 (11.8) | 57.9 (13.2) | 59.0 (11.3)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.982, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Fatigue T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -0.44, 95% CI 2-sided [-6.04 to 5.17] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -4.7 (-8.3, -1.1)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.982, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 1]; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-6.22 to 4.50] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -4.7 (-8.3, -1.1)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.982, Mixed Models Analysis — [p-value comment as in outcome 27, analysis 1]; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-6.32 to 4.36] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 mean change from baseline and 95% confidence interval for the Placebo group was -4.7 (-8.3, -1.1)

28. Secondary Outcome: Change in Baseline in PROMIS - Sleep Disturbance T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Sleep Disturbance T-Score will be used to assess trends over time in this health measure. The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents worse symptomology for the Sleep Disturbance domain. The change from baseline in PROMIS Sleep Disturbance Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1 | 58.6 (7.9) | 56.4 (10.4) | 57.9 (9.1) | 62.6 (7.9)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 56.6 (7.6) | 54.5 (8.7) | 57.7 (8.0) | 57.2 (6.7)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 56.0 (9.7) | 53.7 (6.6) | 56.4 (7.6) | 57.7 (8.6)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 55.4 (9.1) | 56.4 (10.1) | 56.3 (7.6) | 57.2 (8.2)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.607, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Sleep Disturbance T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-4.74 to 4.91] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -3.5 (-6.8, -0.3)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.607, Mixed Models Analysis — [p-value comment as in outcome 28, analysis 1]; Mean Difference (Final Values) = 2.93, 95% CI 2-sided [-1.85 to 7.71] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -3.5 (-6.8, -0.3)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.607, Mixed Models Analysis — [p-value comment as in outcome 28, analysis 1]; Mean Difference (Final Values) = 1.44, 95% CI 2-sided [-3.22 to 6.09] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -3.5 (-6.8, -0.3)

29. Secondary Outcome: Change in Baseline in PROMIS - Social Role Satisfaction T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Social Role Satisfaction T-Score will be used to assess trends over time in this health measure. The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score better functioning for the Social Role Satisfaction domain. The change from baseline in PROMIS Social Role Satisfaction Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1 | 42.2 (5.7) | 42.5 (10.0) | 44.3 (7.3) | 42.4 (7.0)
  Day 29: number analyzed (Participants) | 21 | 24 | 24 | 25
  Day 29 | 44.9 (10.2) | 44.9 (10.7) | 45.1 (9.4) | 47.3 (11.4)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 44.2 (8.1) | 47.1 (9.2) | 47.0 (7.5) | 45.9 (10.3)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 46.1 (9.2) | 48.2 (10.1) | 47.8 (7.7) | 46.8 (9.9)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.981, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Social Role Satisfaction T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-4.66 to 4.30] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 4.2 (0.8, 7.6)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.981, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-3.84 to 4.86] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 4.2 (0.8, 7.6)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.981, Mixed Models Analysis — [p-value comment as in outcome 29, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-4.62 to 4.08] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 4.2 (0.8, 7.6)

30. Secondary Outcome: Change in Baseline in PROMIS - Pain Interference T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Pain Interference T-Score will be used to assess trends over time in this health measure. The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents worse symptomology for the Pain Interference domain. The change from baseline in PROMIS Pain Interference Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/Day 1 | 64.9 (4.9) | 64.7 (7.4) | 65.0 (7.2) | 66.1 (6.4)
  Day 29: number analyzed (Participants) | 21 | 24 | 24 | 25
  Day 29 | 61.6 (7.7) | 61.6 (8.5) | 60.4 (8.9) | 61.2 (10.9)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 61.1 (9.4) | 58.5 (11.2) | 57.7 (7.9) | 62.0 (10.3)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 58.5 (10.2) | 60.4 (6.3) | 60.0 (6.8) | 61.1 (7.4)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.653, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Pain Interference T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -1.85, 95% CI 2-sided [-6.00 to 2.29] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -4.9 (-7.6, -2.1)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.653, Mixed Models Analysis — [p-value comment as in outcome 30, analysis 1]; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-3.10 to 4.88] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -4.9 (-7.6, -2.1)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.653, Mixed Models Analysis — [p-value comment as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-4.31 to 3.67] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -4.9 (-7.6, -2.1)

31. Secondary Outcome: Change in Baseline in PROMIS - Pain Intensity
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Pain Intensity will be used to assess trends over time in this health measure. The Pain Intensity on the PROMIS is a single item numerical rating scale where the respondent selects a whole number representing the average pain of the past 7 days ranging from 0 (no pain) to 10 (worst pain imaginable). The change from baseline in PROMIS Pain Intensity Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Score
  Baseline/ Day 1 | 6.6 (1.4) | 6.9 (1.7) | 7.0 (1.6) | 6.9 (1.7)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 5.5 (2.1) | 5.3 (2.4) | 5.2 (2.6) | 5.8 (2.1)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 5.2 (2.5) | 5.1 (2.8) | 4.9 (2.3) | 5.8 (2.5)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 4.7 (2.2) | 5.2 (2.5) | 4.6 (2.6) | 5.8 (2.3)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.245, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Pain Intensity at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -1.13, 95% CI 2-sided [-2.56 to 0.29] — Estimated mean difference of High JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -1.1 (-2.1, -0.1)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.245, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.93 to 0.80] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -1.1 (-2.1, -0.1)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Test type: Superiority; p = 0.245, Mixed Models Analysis — [p-value comment as in outcome 31, analysis 1]; Mean Difference (Final Values) = -1.28, 95% CI 2-sided [-2.64 to 0.09] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was -1.1 (-2.1, -0.1)

32. Secondary Outcome: Change in Baseline in PROMIS Cognitive Function T-Score
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank version 2.0 - Cognitive Function scale will be used to assess trends over time in this health measure. The raw score is calculated for and translated into a T-score per the PROMIS scoring guide. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation of 10. A higher score represents better cognitive function.
  The change from baseline in PROMIS Cognitive Function Score at Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85) will be assessed.
Time Frame: Visit 1 (Baseline, Day 1), Visit 3 (Day 29), Visit 4 (Day 57), and Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
T-Score
  Baseline/Day 1 | 45.5 (8.5) | 45.1 (9.9) | 42.3 (7.8) | 42.4 (11.0)
  Day 29: number analyzed (Participants) | 21 | 25 | 24 | 25
  Day 29 | 43.6 (9.8) | 48.3 (10.9) | 45.4 (9.2) | 45.4 (12.4)
  Day 57: number analyzed (Participants) | 20 | 23 | 24 | 24
  Day 57 | 44.7 (7.9) | 47.1 (10.9) | 45.6 (9.1) | 43.4 (10.7)
  Day 85: number analyzed (Participants) | 20 | 23 | 23 | 24
  Day 85 | 45.0 (8.5) | 48.1 (10.1) | 45.8 (6.7) | 44.2 (11.2)
Statistical Analysis 1: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.608, Mixed Models Analysis — This p-value is from the overall 3 degree of freedom test that simultaneously compares the mean difference in the change from baseline PROMIS Cognitive Function T-Score at Day 85 for each of the 3 JBT-101 cohorts versus placebo; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-4.45 to 3.54] — Estimated mean difference of High JBT-101 - Placebo in the change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 1.4 (-1.5, 4.4)
Statistical Analysis 2: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.608, Mixed Models Analysis — [p-value comment as in outcome 32, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-2.27 to 5.47] — Estimated mean difference of Medium JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 1.4 (-1.5, 4.4)
Statistical Analysis 3: Comparison: High: JBT-101 20mg/20mg vs Medium: JBT-101 20mg/Placebo vs Low: JBT-101 5mg/5mg vs Placebo; Each active JBT-101 cohort is compared to placebo; Test type: Superiority; p = 0.608, Mixed Models Analysis — [p-value comment as in outcome 32, analysis 1]; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [-2.25 to 5.45] — Estimated mean difference of Low JBT-101 - Placebo in the mean change from baseline at Day 85. The estimated Day 85 change from baseline and 95% confidence interval for the Placebo group was 1.4 (-1.5, 4.4)

33. Secondary Outcome: Percentage of Participants Indicating Clinical Benefit in Treatment Satisfaction
Description: At the end of treatment, the participant and their physician will complete separately a survey asking what treatment assignment they believe they received (e.g., JBT-101, placebo, or cannot tell), whether the participant received benefit from their assigned treatment and whether the participant or their physician would choose the treatment received.
  The percentage of participants who responded that they received clinical benefit from the experimental drug treatment at the end of treatment will be assessed.
Time Frame: Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 22 | 25 | 23 | 23
Percentage of Participants | 59.1 | 76.0 | 69.6 | 52.2

34. Secondary Outcome: Percentage of Physicians Indicating Participant Clinical Benefit in Treatment Satisfaction
Description: At the end of treatment, the participant and their physician will complete separately a survey asking what treatment assignment they believe they received (e.g., JBT-101, placebo, or cannot tell), whether the participant received benefit from their assigned treatment and whether the participant or their physician would choose the treatment received.
  The percentage of physicians who responded that the participant received clinical benefit from the experimental drug treatment at the end of treatment will be assessed.
Time Frame: Visit 5 (Day 85 - Last Day of Treatment)
Population: as for outcome 12
Measure: Number; unit: Percentage of Physicians
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 23 | 25 | 23 | 24
Percentage of Physicians | 43.5 | 60.0 | 65.2 | 66.7

35. Secondary Outcome: Number of Grade 3 or Higher Treatment-emergent Adverse Events (TEAE) Related to Study Product
Description: Treatment-emergent Adverse Events grading will be defined by the National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. The number of TEAE will be identified by monitoring participant-reported AEs, vital signs, medical history, physical exams, blood and urine safety tests, 12-lead electrocardiograms, and the Addiction Research Center Inventory-Marijuana (ARCI-M). TEAE are defined as AEs that, in the opinion of the blinded/masked site investigator, are " possibly", "probably" or "definitely" related to the assigned study treatment.
Time Frame: Day 1 after initiation of study intervention through Day 113
Population: The safety population includes all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Events
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Number of Events | 1 | 0 | 0 | 0

36. Secondary Outcome: Number of Treatment Emergent QTc Prolongation Events
Description: The number of treatment emergent QTc prolongation events will be identified when QTc prolongation > 500 msec total duration and when the change from Visit 1 (Day 1) QTc interval prior to study drug administration > 60 msec Twelve-lead ECGs were recorded in triplicate at Screening and Visits 1 (Day 1) and 5 (Day 85). The ECGs were evaluated for medically significant abnormalities and QT/QTc intervals. The QT/QTc intervals were measured at Visit 1 (Day 1) before administration and between 2.5 and 3.5 hours after administration of study product in the clinic, at the time of maximum JBT-101 concentration in the blood.
Time Frame: Visit 1 (Baseline, Day 1) and Visit 5 (Day 85 - Last Day of Treatment)
Population: The safety population includes all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Events
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Number of Events | 0 | 0 | 0 | 0

37. Secondary Outcome: Number of SLE Disease Flares by Severity Using the SELENA-SLEDAI Flare Index (SFI)
Description: The number of mild/moderate and severe disease flares will be assessed using the SFI instrument to define disease flare(s) and severity.
  The SELENA SLEDAI Flare Index categorizes disease flares as mild/moderate or severe, based on the highest categories of clinical features recorded or by treatment recommendations by the physician.
Time Frame: Visit 3 (Day 29)
Population: The safety population includes all participants who received at least one dose of study treatment. Number of participants analyzed is number of participants in the safety population with data at the visit.
Measure: Number; unit: Number of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 21 | 25 | 24 | 25
Number of Participants
  Severe | 1 | 1 | 1 | 0
  Mild/Moderate | 4 | 2 | 0 | 3
  No Flare | 16 | 22 | 23 | 22

38. Secondary Outcome: Number of SLE Disease Flares by Severity Using the SELENA-SLEDAI Flare Index (SFI)
Description: as for outcome 37
Time Frame: Visit 4 (Day 57)
Population: as for outcome 37
Measure: Number; unit: participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 24 | 24
participants
  Severe | 1 | 0 | 0 | 0
  Mild/Moderate | 2 | 3 | 3 | 7
  No Flare | 17 | 20 | 21 | 17

39. Secondary Outcome: Number of SLE Disease Flares by Severity Using the SELENA-SLEDAI Flare Index (SFI)
Description: as for outcome 37
Time Frame: Visit 5 (Day 85)
Population: as for outcome 37
Measure: Number; unit: participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 23 | 24
participants
  Severe | 0 | 1 | 2 | 1
  Mild/Moderate | 3 | 4 | 2 | 4
  No Flare | 17 | 18 | 19 | 19

40. Secondary Outcome: Number of SLE Disease Flares by Severity Using the SELENA-SLEDAI Flare Index (SFI)
Description: as for outcome 37
Time Frame: Visit 6 (Day 113)
Population: as for outcome 37
Measure: Number; unit: participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 23 | 24
participants
  Severe | 0 | 0 | 0 | 2
  Mild/Moderate | 7 | 5 | 9 | 9
  No Flare | 13 | 18 | 14 | 13

41. Secondary Outcome: Number of BILAG-2004 Disease Flares
Description: The number of BILAG-2004 disease flares as defined as one new BILAG A or two new BILAG B scores will be assessed.
  The BILAG-2004* is a validated index for assessing SLE disease activity. The BILAG-2004 includes 97 clinical and laboratory items to evaluate SLE disease activity in 9 organ systems.
  * BILAG-2004: British Isles Lupus Assessment Group 2004.
Time Frame: Visit 3 (Day 29)
Population: as for outcome 37
Measure: Number; unit: Number of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 21 | 25 | 24 | 25
Number of Participants
  One new BILAG A Flare | 0 | 0 | 0 | 0
  Two new BILAG B Flares | 0 | 1 | 0 | 0

42. Secondary Outcome: Number of BILAG-2004 Disease Flares
Description: as for outcome 41
Time Frame: Visit 4 (Day 57)
Population: as for outcome 37
Measure: Number; unit: Number of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 24 | 24
Number of Participants
  One new BILAG A Flare | 0 | 0 | 0 | 1
  Two new BILAG B Flares | 0 | 0 | 1 | 0

43. Secondary Outcome: Number of BILAG-2004 Disease Flares
Description: as for outcome 41
Time Frame: Visit 5 (Day 85)
Population: as for outcome 37
Measure: Number; unit: Number of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 23 | 24
Number of Participants
  One new BILAG A Flare | 2 | 0 | 0 | 1
  Two new BILAG B Flares | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of BILAG-2004 Disease Flares
Description: as for outcome 41
Time Frame: Visit 6 (Day 113)
Population: as for outcome 37
Measure: Number; unit: Number of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 20 | 23 | 23 | 24
Number of Participants
  One new BILAG A Flare | 0 | 0 | 1 | 0
  Two new BILAG B Flares | 1 | 0 | 0 | 0

45. Secondary Outcome: Number of Treatment Emergent Events With Elevated Liver Tests
Description: The number of participants with elevated liver tests, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 x upper limit of normal and total bilirubin > 1.5 x the upper limit of normal, present on repeat testing, at Visit 3 (Day 29), Visit 4 (Day 57), Visit 5 (Day 85) and Visit 6 (Day 113) will be assessed.
Time Frame: Day 1 through Visit 6 (Day 113)
Population: The safety population includes all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Events
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Number of Events | 0 | 0 | 0 | 0

46. Secondary Outcome: Number of Treatment Emergent Intolerability Events
Description: The number of intolerability events of the study drug, defined as incidence of discontinuation of study product due to TEAEs at least possibly related to study product from Visits 1 (Day 1) through 5 (Day 85) will be assessed.
Time Frame: Day 1 after initiation of study intervention through Visit 5 (Day 85 - Last Day of Treatment)
Population: The safety population includes all participants who received at least one dose of study treatment.
Measure: Number; unit: Number of Events
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Number of Events | 6 | 4 | 0 | 0

47. Secondary Outcome: Percentage of Participants With Increased Scores From Baseline on ARCI-M
Description: The percentage of participants who experienced ≥1 score increase on the ARCI-M from the Visit 1 (Day 1) pre-dose assessment at Visit 1 (Day 1) post-dose, Visit 3 (Day 29) and Visit 5 (Day 85) will be assessed.
  The ARCI-M questionnaire was completed by subjects at Visit1 (Day 1) pre- and post-dosing, Visit 3 (Day 29) and Visit 5 (Day 85). This is a 12-item true/false questionnaire developed by the National Institutes of Drug Abuse, designed to detect the full range of subjective responses experienced by marijuana users. An answer of true has an assigned value of 1 and an answer of false has an assigned value of 0. The ARCI-M score was computed as the sum of the assigned values for all 12 questions and can range from 0 to 12. If a question is missed, the score is not calculated.
Time Frame: Visit 1 (Baseline, Day 1-prior to treatment initiation), Visit 1 (Baseline, Day 1-post-treatment initiation) Visit 3 (Day 29) and Visit 5 (Day 85 - Last Day of Treatment)
Population: mITT
Measure: Number; unit: Percentage of Participants
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
Number analyzed (Participants) | 25 | 27 | 24 | 25
Percentage of Participants
  Day 1 Post-Dose: number analyzed (Participants) | 24 | 27 | 24 | 25
  Day 1 Post-Dose | 25.0 | 11.1 | 20.8 | 4.0
  Day 29: number analyzed (Participants) | 20 | 24 | 24 | 25
  Day 29 | 45.0 | 37.5 | 29.2 | 36.0
  Day 85: number analyzed (Participants) | 18 | 23 | 22 | 23
  Day 85 | 11.1 | 39.1 | 27.3 | 56.5

ADVERSE EVENTS:
Time Frame: AEs of Grade 2 and above will be collected from time of signing of informed consent until the participant completes study participation, or until 30 days after he/she prematurely withdraws (without withdrawing consent), or is withdrawn from the study, up to 20 weeks.
Description: National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Arm/Group | High: JBT-101 20mg/20mg | Medium: JBT-101 20mg/Placebo | Low: JBT-101 5mg/5mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 3/27 | 0/24 | 2/25
Other Adverse Events (participants affected / at risk) | 10/25 | 11/27 | 16/24 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High: JBT-101 20mg/20mg (N=25) | Medium: JBT-101 20mg/Placebo (N=27) | Low: JBT-101 5mg/5mg (N=24) | Placebo (N=25)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Serositis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High: JBT-101 20mg/20mg (N=25) | Medium: JBT-101 20mg/Placebo (N=27) | Low: JBT-101 5mg/5mg (N=24) | Placebo (N=25)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 7 (11) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 3 (4) | 4 (4) | 1 (1) | 5 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 2 (2) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT03093402/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT03093402/SAP_001.pdf